CLINICAL TRIAL: NCT04863326
Title: Evaluation of the Making Proud Choices! Teen Pregnancy Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Office of Population Affairs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHSP23337014T
Record Dates: First submitted 2021-04-20; First posted 2021-04-28 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Teen Pregnancy Prevention
MeSH Terms: interventions — Commerce

STUDY DESIGN:
Intervention Model Description: The MPC curriculum aims to provide adolescents with the information and tools they need to reduce their risk of sexually transmitted diseases (STDs), HIV, and pregnancy. The curriculum emphasizes abstinence as the safest choice for avoiding pregnancy and STDs, but also encourages youth to use condoms and other methods of birth control if they do have sex. The curriculum includes video clips, student role-playing activities, and group discussions. It also involves skill-building activities for correct condom use, refusal techniques, and safer-sex negotiation, and opportunities for students to practice these skills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Making Proud Choices (Experimental): This evaluation tests the effect of the MPC School Edition, the version of the MPC 5th Edition designed for implementation in school. This edition includes 9.5 hours of content implemented in 14 40-minute modules. Schools assigned to the MPC condition received MPC in a targeted class.
  Interventions: Behavioral: Making Proud Choices
- Business as usual (Active Comparator): The control group continued with their regular programming in the targeted class, which was often a health or Reserve Officer Training Corps (ROTC) class.
  Interventions: Behavioral: Business as usual

INTERVENTIONS:
Behavioral: Making Proud Choices
  Arms: Making Proud Choices
Behavioral: Business as usual
  Arms: Business as usual

SUMMARY:
Under contract to the Office of Population Affairs (OPA), Mathematica is conducting an impact study of the Making Proud Choices! (MPC) teen pregnancy prevention program. The impact study is designed to estimate the impact of MPC, compared to the business-as-usual condition, on risk and protective factors, sexual behaviors, and longer term health goals including pregnancy and sexually transmitted infections.

DETAILED DESCRIPTION:
This evaluation used a cluster randomized controlled trial (RCT) design to assess the effectiveness of MPC, with schools within districts randomly assigned to one of two conditions: (1) MPC implemented by health educators, or (2) business as usual. In total, 31 school clusters were randomly assigned to condition, including roughly 2800 students, in four geographic areas across the U.S.

The study was implemented over the course of three school years (2016-17, 2017-18 and 2018-19), with youth in each year considered a separate evaluation cohort, and with participating schools (and new cohorts of eligible youth) randomized to condition each year.

There are two main sources of data for this study: outcome and implementation data. Youth in the study completed two waves of self-report surveys: (1) a baseline survey administered before programming began, and (2) a follow-up outcome survey administered approximately six months after the end of programming (approximately 9 months after baseline, on average). The surveys measured antecedents to sexual behavior (risk and protective factors), sexual behaviors, and ultimately, MPC's health goals of reducing sexually transmitted infections and teen pregnancies. Program implementation data included fidelity and attendance logs, observations, interviews, study youth focus groups, staff surveys, and technical assistance logs.

The benchmark analytic approach for estimating program impacts focuses on individuals with observed (non-missing) outcome data, and will statistically adjust for several baseline and location variables to produce credible and precise estimates of program effectiveness. Several sensitivity analyses will be conducted to understand the robustness of the findings across alternative specifications, and to understand the effect of MPC across a variety of subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a study school
* Attending the targeted class (e.g. health class) for the first time

Exclusion Criteria:

* None

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2810 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Knowledge about HIV | Survey administered 6 months post program
  Proportion of knowledge items about HIV/STDs answered correctly.
Knowledge about pregnancy | Survey administered 6 months post program
  Proportion of knowledge items about pregnancy answered correctly.
Knowledge about condoms | Survey administered 6 months post program
  Proportion of knowledge items about condom use answered correctly.
Knowledge about other forms of contraception | Survey administered 6 months post program
  Proportion of knowledge items about contraceptive use answered correctly.
Belief that sex may adversely affect future goals | Survey administered 6 months post program
  Proportion of statements about how sexual activity will interfere with goals and dreams that the respondent agrees or strongly agrees with.
Belief that condoms can be pleasurable | Survey administered 6 months post program
  Proportion of statements about how condoms can be pleasurable that the respondent agrees or strongly agrees with.
Attitudes about condoms | Survey administered 6 months post program
  Proportion of statements about condom use that the respondent either agrees or strongly agrees with.
Condom self-efficacy | Survey administered 6 months post program
  Proportion of statements about self-efficacy using condoms that the respondent agrees or strongly agrees with.
Condom negotiation | Survey administered 6 months post program
  Proportion of statements about self-efficacy negotiating condom that the respondent agrees or strongly agrees with.
Refusal skills | Survey administered 6 months post program
  Proportion of statements about self-efficacy refusing sex with a partner that the respondent agrees or strongly agrees with.
Ever any sex (vaginal, oral, or anal) | Survey administered 6 months post program
  Binary variable representing if the respondent reported having ever had vaginal, oral, or anal sex.
Any sex (in past 3 months) | Survey administered 6 months post program
  Binary variable representing if the respondent reported having vaginal, oral, or anal sex in the three month period before completing the follow-up survey.
Times having any sex (in past 3 months) | Survey administered 6 months post program
  Count variable representing the total number of times respondent had vaginal, oral and/or anal sex in the three month period before completing the follow-up survey.
Count of vaginal sex partners (in the past 3 months) | Survey administered 6 months post program
  Count variable representing the number of partners for vaginal sex in the three month period before completing the follow-up survey.
Any sex without a condom (in past 3 months) | Survey administered 6 months post program
  Binary variable representing if respondent reported having any risk for STD/STI sex (sex without a condom) in the three month period before completing the follow-up survey.
Times having any sex without a condom in past 3 months | Survey administered 6 months post program
  Count variable representing the total number of times respondent had risky sex in the three months before completing follow-up survey.
Sex without birth control in past 3 months | Survey administered 6 months post program
  Binary variable representing if respondent reported having had unprotected vaginal sex in the three months before completing the follow-up survey.
Times having sex without birth control (in past 3 months) | Survey administered 6 months post program
  Count variable representing the total number of times the respondent had unprotected vaginal sex in the three month period before completing the follow-up survey.
Ever pregnant | Survey administered 6 months post program
  Binary variable representing if the respondent reported a pregnancy or has gotten someone pregnant.
Any sexually transmitted infection (STI) | Survey administered 6 months post program
  Binary variable representing if the respondent indicated having been told they have a sexually transmitted infection.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cole R, Neelan TS, Langan A, Keating B, Walzer J, Asheer S, Zief S. The Impact of Making Proud Choices! on Youth's Sexual Health Attitudes, Knowledge, and Behaviors. J Adolesc Health. 2024 Apr;74(4):787-793. doi: 10.1016/j.jadohealth.2023.10.031. Epub 2023 Dec 13. PMID 38099897